CLINICAL TRIAL: NCT02896881
Title: Interest of New MRI Sequences After Embolization of Brain Arteriovenous Malformations (MAV-IRM)
Brief Title: Interest of New MRI Sequences After Embolization of Brain Arteriovenous Malformations
Acronym: MAV-IRM
Status: Terminated | Type: Observational
Why Stopped: The study no longer recruits patients, and its scientific relevance to healthcare practice has become obsolete.
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: RBC_2016_7
Record Dates: First submitted 2016-09-07; First posted 2016-09-12 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Brain Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In previous studies exploring specific sequences of MRI (susceptibility weighted imaging (SWI) and arterial spin labeling (ASL)), the investigators have shown the great sensibility of these MRI sequences to detect arteriovenous shunts, compared to angiography imaging (static or dynamic). This prospective study aims to compare multisequence MRI to brain arteriography imaging in patients undergoing brain arteriovenous malformations embolization.

DETAILED DESCRIPTION:
Cerebral arteriovenous malformations are treated to eliminate the potential risk of haemorrhage. There are three possible treatment modalities: surgery, radiosurgery or embolisation. Complete exclusion of the arteriovenous malformation is a prerequisite for confirming that there is no residual risk of haemorrhage. After treatment, arteriography is the gold standard for confirming this exclusion. The absence of early opacification of the venous drainage is considered a sign of cure.

Several arteriographic aspects are possible after treatment by embolisation:

* Arteriography may be strictly normal (no abnormalities).
* The persistence of early venous opacification (presence of arterialised blood) indicates the persistence of a residual AVM.
* Other vascular anomalies without early venous drainage may be present: dysplastic vessels (irregular shape, "corkscrew" appearance) ; capillary blush in the embolisation bed (hyperaemia) ; other: slow flow, slow filling, or widening of afferent arteries.

Our previous studies exploring the use of specific MRI sequences, in magnetic susceptibility (SWI), arterial spin labelling (ASL) and angiography (static or dynamic) sequences, have enabled us to demonstrate the very high sensitivity of these sequences for detecting an arteriovenous shunt, whether native (when the AVM is discovered) or residual after treatment. We would like to carry out a prospective study to compare cerebral arteriography and MRI (multi-sequence) in patients treated by embolisation for cerebral arteriovenous malformation.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* with brain Arteriovenous Malformations
* embolization treatment scheduled

Exclusion Criteria:

* patient's refusal to participate in the study
* contraindication to undergo MRI examination
* patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with brain Arteriovenous Malformations and embolization treatment scheduled.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
sensitivity of multisequence MRI to detect a residual arteriovenous malformation after embolization | within 3 months after embolization
  Early opacification of a vein, possibly associated with the presence of abnormal vessels, will be sought, indicating a residual malformation. After interpretation of the MRI (angio-MRI with multi-sequences, magnetic susceptibility (SWI), arterial spin labelling (ASL) and static or dynamic angiography), the result will be coded dichotomously: (presence/absence of a residual malformation). The arteriography result will be coded in the same way. The sensitivity of the new MRI sequences for detecting a residual arteriovenous malformation after treatment by embolisation will thus be assessed, compared with arteriography (gold-standard).

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël BLANC, MD, Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild
Locations (1):
- Fondation Opthalmologique A de Rothschild, Paris, France